CLINICAL TRIAL: NCT00906451
Title: Phase 4 Study of the Effect of Simvastatin Treatment on Inflammatory Response and Endothelial Function After Myocardial Infarction
Brief Title: Simvastatin Effect on Inflammation and Endothelial Function After Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia Heart Study Group (Other)
Responsible Party: Andrei C. Sposito, University of Brasilia Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Simvastatin Post-MI
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-05

CONDITIONS: Myocardial Infarction; Inflammation; Endothelial Dysfunction
Keywords: myocardial infarction; inflammation; endothelial dysfunction
MeSH Terms: conditions — Myocardial Infarction; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No lipid-lowering (No Intervention): No lipid-lowering treatment during the first 7 days and then simvastatin 20 mg/day for three additional weeks, till the endothelial function assessment
  Interventions: Drug: Simvastatin
- Simvastatin 20 mg (Experimental): Simvastatin 20 mg/day for 30 days, till the endothelial function assessment
  Interventions: Drug: Simvastatin
- Simvastatin 40 mg (Experimental): Simvastatin 40 mg/day for 7 days and then switched to simvastatin 20mg/day for additional 3 weeks, till the endothelial function assessment
  Interventions: Drug: Simvastatin
- Simvastatin 80 mg (Experimental): Simvastatin 80 mg/day for 7 days and then switched to simvastatin 20 mg/day for additional 3 weeks, till the endothelial function assessment
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin

SUMMARY:
During myocardial infarction, inflammatory response may negatively influence ventricle wall remodeling as well as endothelium-dependent vasomotor function in the coronary and systemic arterial systems. Statins have been consistently proved to attenuate inflammation and improve endothelial function. In this study, we tested the effect of different doses of statin on inflammatory response and endothelium-dependent vasodilation.

DETAILED DESCRIPTION:
During acute coronary syndromes (ACS), the generation of inflammatory mediators negatively influences arterial wall remodeling and the endothelium-dependent vasomotor function in the coronary and systemic arterial systems. The intensity of this inflammatory upregulation is strongly related to the incidence of recurrent coronary events. High dose potent statins can rapidly reduce plasma levels of cholesterol-rich lipoproteins and inflammatory activity in subjects during ACS. By inference, it is plausible to hypothesize that these effects during the acute phase of myocardial infarction may influence the post-discharge endothelial dysfunction. So far, data is unavailable to verify this assumption or to define the potency required for such statin anti-inflammatory effect in myocardial infarction patients. The present study aim to investigate the role of statin dose on the time-course of the inflammatory response during the acute phase of myocardial infarction and its late effect on endothelium-dependent arterial dilation.

ELIGIBILITY:
Inclusion Criteria:

* Less than 24 hours after the onset of MI symptoms
* ST-segment elevation of a least 1 mm (frontal plane) or 2 mm (horizontal plane) in two contiguous leads
* Myocardial necrosis, as evidenced by increased CK-MB and troponin levels

Exclusion Criteria:

* Use of statins for at least 6 months prior the myocardial infarction

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Elevation of plasma C reactive protein | Five days
  Changes in CRP levels between the first and fifth day after myocardial infarction

SECONDARY OUTCOMES:
Brachial Artery Endothelial function | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, MD, PhD, Study Chair — University of Brasilia Medical School
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Result] Sposito AC, Santos SN, de Faria EC, Abdalla DS, da Silva LP, Soares AA, Japiassu AV, Quinaglia e Silva JC, Ramires JA, Coelho OR. Timing and dose of statin therapy define its impact on inflammatory and endothelial responses during myocardial infarction. Arterioscler Thromb Vasc Biol. 2011 May;31(5):1240-6. doi: 10.1161/ATVBAHA.110.218685. Epub 2011 Mar 3. PMID 21372302